CLINICAL TRIAL: NCT04526366
Title: Apnoea-Hypopnoea-Indices Determined Via Continuous Posi-tive Airway Pressure (AHI-CPAPflow) Versus Those Determined by Polysomnography (AHI-PSGgold): a Protocol for a Systematic Review and Meta-analysis
Brief Title: Apnoea-Hypopnoea-Indices Determined Via Continuous Positive Airway Pressure vs Those Determined by Polysomnography
Acronym: Meta IAHflow
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0395
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Sleep Apnea Syndromes
Keywords: apnoea hypopnoea index; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure; Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: All (full scientific) study designs and publication types written in English and reporting Bland-Altman test results (or other tests suggesting the presence of the required data) between simultaneous, paired, polysomnography (PSG)-derived AND Continuous Positive Airway Pressure (CPAP)-derived data describing sleep disordered breathing.
  Interventions: Device: Continuous Positive Airway Pressure; Device: Polysomnography

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure device deployed for at least one night synchronously with polysomnography.
Device: Polysomnography — Polysomnography deployed for at least one night synchronously with Continuous Positive Airway Pressure.

SUMMARY:
To date, no published systematic review and meta-analysis has compared AHI-CPAPflow and AHI-PSGgold. Therefore, the primary objective of this study is to compare published data for AHI-PSGgold and AHI-CPAPflow in patients treated by CPAP.

DETAILED DESCRIPTION:
The secondary objectives are to evaluate, in a manner similar to the primary objective, data for apnoea indices (AI), hypopnoea indices (HI), respiratory disturbance indices (RDI) and respiratory effort related arousals (RERAs) and to perform subgroup analyses focusing on the inclusion/exclusion of central apnoea patients, BMI levels, CPAP device brands, pressure titration modes, use of a predetermined and fixed pressure level or not, and the impact of a 4%-PSG desaturation criteria versus 3%-PSG on index accuracy.

ELIGIBILITY:
Inclusion Criteria:

* All (full scientific) study designs and publication types written in English and reporting Bland-Altman test results (or other tests suggesting the presence of the required data) between simultaneous, paired, polysomnography (PSG)-derived AND Continuous Positive Airway Pressure (CPAP)-derived data describing sleep disordered breathing.

Exclusion Criteria:

* Duplicates
* Does not refer to a full scientific article (e.g. case reports are excluded).
* Meta-analysis
* Paediatric populations (populations <18 years are excluded).
* Absence of appropriate paired results: synchronized polysomnography (PSG)-derived AND Continuous Positive Airway Pressure (CPAP)-derived data must be reported for ≥1 of the following measures: Apnoea-Hypopnoea-Indices (AHI), Apnoea-Indices (AI), Hypopnoea-Indices(HI), respiratory disturbance index (RDI), respiratory effort related arousals (RERA).
* Absence of appropriate test comparing paired results: the study must use ≥1 of the fol-lowing tests to compare the previously mentioned PSG-vs-CPAP-derived data: a bland-altman or correlation test, other conformity tests, tests of differences in centrality.
* Inappropriate PSG scoring 1: PSG-derived variables must be coded following the American Academy of Sleep Medicine 2007 (or more recent) guidelines.
* Inappropriate PSG scoring 2: PSG-derived variables must be scored manually.
* Inappropriate PSG scoring 3: oxygen desaturation level used for scoring must be mentioned and at 3% or 4%.
* Inappropriate CPAP description: brand/device names must be mentioned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with a CPAP-device and synchronous polysomnography.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
The mean difference between AHI-CPAPflow and AHI-PSGgold | Day 0
  AHI-CPAPflow = Apnoea-Hypopnoea-Indices Determined Via Continuous Positive Airway Pressure AHI-PSGgold = Apnoea-Hypopnoea-Indices Determined by Polysomnography
The standard deviation for the mean difference between AHI-CPAPflow and AHI-PSGgold | Day 0

SECONDARY OUTCOMES:
The mean difference between AI-CPAPflow and AI-PSGgold | Day 0
  AI-CPAPflow = Apnoea--Indices Determined Via Continuous Positive Airway Pressure AI-PSGgold = Apnoea--Indices Determined by Polysomnography
The standard deviation for the mean difference between AI-CPAPflow and AI-PSGgold | Day 0
The mean difference between HI-CPAPflow and HI-PSGgold | Day 0
  HI-CPAPflow = Hypopnoea--Indices Determined Via Continuous Positive Airway Pressure HI-PSGgold = Hypopnoea--Indices Determined by Polysomnography
The standard deviation for the mean difference between HI-CPAPflow and HI-PSGgold | Day 0
The mean difference between RDI-CPAPflow and RDI-PSGgold | Day 0
  RDI-CPAPflow = Respiratory Disturbance Indices Determined Via Continuous Positive Airway Pressure RDI-PSGgold = Respiratory Disturbance Indices Determined by Polysomnography
The standard deviation for the mean difference between RDI-CPAPflow and RDI-PSGgold | Day 0
The mean difference between RERA-CPAPflow and RERA-PSGgold | Day 0
  RERA-CPAPflow = Respiratory Effort Related Arousals Determined Via Continuous Positive Airway Pressure RERA-PSGgold = Respiratory Effort Related Arousals Determined by Polysomnography
The standard deviation for the mean difference between RERA-CPAPflow and RERA-PSGgold | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Dany Jaffuel, MD,PhD, Study Director — University Hospitals of Montpellier
Locations (1):
- University Hospitals of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertelli F, Suehs CM, Mallet JP, Rotty MC, Pepin JL, Gagnadoux F, Matzner-Lober E, Bourdin A, Molinari N, Jaffuel D. Apnoea-hypopnoea indices determined via continuous positive airway pressure (AHI-CPAPflow) versus those determined by polysomnography (AHI-PSGgold): a protocol for a systematic review and meta-analysis. BMJ Open. 2021 May 10;11(5):e044499. doi: 10.1136/bmjopen-2020-044499. PMID 33972338
- See also: Meta IAHflow on the Open Science Framework. — https://osf.io/gycw2/